CLINICAL TRIAL: NCT06588049
Title: Nitrate Mouth Rinse and the Oral Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Leigha Rock, Director - School of Dental Hygiene, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-7166
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-09

CONDITIONS: Nitric Oxide; Oral Microbiome
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate Mouth Rinse (Experimental): Nitrate suspension with approximately 50-100mg nitrates formulated with water swished in mouth for 30 seconds and then expectorated once daily for 14 consecutive days.
  Interventions: Dietary Supplement: Beet Root
- Water Mouth Rinse (Placebo Comparator): Water mouth rinse swished in mouth for 30 seconds and then expectorated once daily for 14 consecutive days.
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Beet Root — Beet Root powder used as a mouth rinse in suspension with water
  Arms: Nitrate Mouth Rinse
Other: Water — Water used as a mouth rinse
  Arms: Water Mouth Rinse

SUMMARY:
The study is aimed to determine if changes to the oral microbiome occur after the use of a nitrate rich mouth rinse. Participants with be asked to use either a controlled (water) mouthrinse once daily for 2 weeks while maintaining normal oral hygiene practices, or use the nitrate rich mouthrinse once daily for 2 weeks.

Primary Outcome measures:

-changes in the composition of the oral microbiome

Secondary Outcome measures

* Blood Pressure
* Salivary Nitric Oxide Levels

DETAILED DESCRIPTION:
Nitrate is found in high concentrations in beet root, and as such we will use a beet root based product as a daily mouth rinse (Swish and Spit) as a part of the participants daily oral hygiene regimen and collect the participants biofilm before and after 2 weeks of regular use. We will then analyze the data using 16s rRNA sequencing to evaluate the changes in alpha diversity, beta diversity and the absolute and relative differential abundance of nitrate reducing bacteria in the oral microbiome. We will also collect salivary samples to evaluate NO levels, as well as measure blood pressure pre and post treatment.

After this study's completion, we expect to have gained new knowledge on nitrate's influence on the oral microbiome's composition. Gaining this knowledge will allow better public understanding of the effects oral hygiene products have on their oral and systemic health. In addition, the knowledge gained could encourage further investigations into how to better formulate oral hygiene products for improved health and performance.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 18 and 40. Have no uncontrolled systemic diseases.

Participants with mild chronic conditions such as:

* Asthma
* Type 1 Diabetes Mellitus

Exclusion Criteria:

* You are under the age of 18.
* You have uncontrolled systemic diseases, or acute infections.
* You are taking prescription, antibiotics, probiotics, or antimicrobial mouthrinses.
* You have a documented true allergy (i.e Hives, Swelling of lips/throat) Soy, Nuts, Seeds, Dairy, Egg products, Fish/Shellfish or Wheat.
* The presence of acute or chronic oral conditions including:

  * Herpes Simplex Virus (recent cold sores)
  * Stomatitis
  * Oral Lichen Planus
  * Angular Cheilitis
  * Candidiasis
  * Necrotizing Gingival Diseases
  * Other inflammatory or infectious pathologies
  * Active dental caries "cavities"
  * Any other periodontal diagnosis other than 'Healthy Periodontium' or localized gingivitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Microbial composition | 2 weeks
  16s rRNA sequencing will be used to explore alpha and beta diversity pre- and post-intervention. Absolute and relative differential abundance will be examined. Functional prediction analysis will be explored.

SECONDARY OUTCOMES:
Blood Pressure | 2 weeks
  Systolic and diastolic pressures
Nitric Oxide | 2 weeks
  Salivary samples will be obtained to determine Nitric Oxide levels

CONTACTS AND LOCATIONS:
Overall Officials: Leigha Rock, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
deidentifed data and sequencing will be uploaded to a public repository such as the Gene Expression Omnibus.